CLINICAL TRIAL: NCT01757041
Title: The Clinical and Molecular Epidemiology of Streptococcus Agalactiae (Group B Streptococcus)Maternal Colonisation and Association With Adverse Perinatal Outcomes
Brief Title: The Clinical and Molecular Epidemiology of Streptococcus Agalactiae Colonisation on the Kenyan Coast
Acronym: GBS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: B9RUHL0
Record Dates: First submitted 2012-11-28; First posted 2012-12-28 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Streptococcus Agalactiae (Streptococcus Group B)
Keywords: Streptococcus agalactiae; Maternal; Newborn; Africa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sub-Saharan Africa (sSA) has the highest regional rates of perinatal mortality worldwide. Group B Streptococcus (GBS) has been identified as a leading cause of early onset neonatal sepsis (EOS, in <7 days of life) in sSA. In other regions, maternal carriage is associated with early onset neonatal sepsis, but in addition, other adverse perinatal outcomes (stillbirths, early neonatal death, low birth weight and prematurity). Robust data on maternal GBS carriage in sSA and its burden on adverse perinatal outcomes are lacking, with important consequences for public health interventions.

Through investigation of maternal carriage and perinatal outcomes at three different sites: rural, semi-rural and urban, this study will provide a comprehensive description of the burden of GBS in coastal Kenya, informing public health policy and driving forward interventions. Risk factors for maternal colonisation and invasive neonatal disease will be assessed, including through retrospective immunological investigation of cord blood in neonates subsequently identified as having invasive GBS disease or other adverse perinatal outcomes, compared to those without.

GBS isolates from maternal colonisation will be typed (sero-typing and molecular analysis), and these isolates will be compared to existing archived neonatal isolates from investigation of neonatal sepsis in KDH (Kilifi District Hospital). This is important so that we know the prevalent sub-types causing neonatal disease in Kenya, those which are carried by mothers, and therefore whether maternal GBS carriage correlates with a high risk of perinatal disease. GBS vaccines in development are type-specific and this will inform their use in sSA.

Stillbirths will also be investigated, in individual cases, through additional detailed microbiological and other laboratory investigations to make an assessment of the contribution of GBS to stillbirths in Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Admitted for delivery

Exclusion Criteria:

* Consent refusal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mothers admitted for delivery to participating health centres (Kilifi District Hospital, Coast Provincial General Hospital, Bamba sub-District Hospital, Ganze Health Facility).
Sampling Method: Probability Sample
Enrollment: 7967 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maternal recto-vaginal GBS colonisation | Single time point (at delivery)
  Prevalence of GBS recto-vaginal carriage in pregnant mothers in rural, semi-rural and urban sites.

SECONDARY OUTCOMES:
Stillbirths | Single time point (at delivery)
  Association of stillbirth with Group B Streptococcus
Neonatal GBS Colonisation | Within 4h of delivery
  Prevalence of neonatal GBS colonization
Preterm birth | Single time point (at delivery)
  Determine association between GBS and preterm birth
Low birth weight | Single time point (at delivery)
  Association of GBS with low birth weight babies

CONTACTS AND LOCATIONS:
Overall Officials: Anna Seale, BMBCh, Principal Investigator — KEMRI-Wellcome Trust and University of Oxford
Locations (4):
- Kenya (4):
  - Bamba sub-District Hospital, Bamba, Coast
  - Ganze Health Facility, Ganze, Coast
  - Kilifi District Hospital, Kilifi, Coast
  - Coast Provincial General Hospital, Mombasa, Coast